CLINICAL TRIAL: NCT02944318
Title: The Movement Program for an Active and Healthy Lifestyle in Adolescents and Its Relationship With School Performance
Brief Title: The Movement Program for an Active and Healthy Lifestyle in Adolescents
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kelly Samara da Silva (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Kelly Samara da Silva, Principal Investigator, Universidade Federal de Santa Catarina
Organization: Universidade Federal de Santa Catarina (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1.259.910
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Adolescent Behavior
Keywords: Physical Activity; Healthy Lifestyle; Academic performance
MeSH Terms: conditions — Adolescent Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "The Movement" Program (Experimental): The intervention program was structured according three main components: (1) training and activities in general curriculum and Physical Education classes; (2) active facilities in the school environment; (3) health education in school community.
  Interventions: Behavioral: The Movement Program
- No intervention (No Intervention): Schools in the control group will maintain a regular academic year with conventional activities. Thus schools have two weekly Physical Education classes which are organized by according to the perspective of their teachers. Besides that, the Program "Saúde na Escola" is also performed.

INTERVENTIONS:
Behavioral: The Movement Program — The program duration will be one academic year (around ten months) in 2017. The intervention strategies will focus on: (1) teachers' training and activities on health in curriculum; (2) active opportunities in the school environment (facilities and materials for PA practice) and (3) health education (posters and folders to students and parents).
  Arms: "The Movement" Program

SUMMARY:
School is a favorable environment for the development of actions aimed at healthy behavioral changes. This project proposes to evaluate the effectiveness of an intervention program on aspects of lifestyle, with a focus on physical activity (PA) and reducing sedentary behaviors, and the relationship of these factors with the academic performance of students in the school from Florianopolis, SC, Brazil.

This is a randomized controlled intervention study enroling classes of 7th to 9th grade of fundamental education.

The intervention program will last for one year (about ten months), with three focuses: training of teachers, educational and environmental changes to behavior change.

ELIGIBILITY:
Inclusion Criteria:

Students of both sexes Students aged 12-15 years Students who are enrolled in 7-9 grade classes

Exclusion Criteria:

Students younger than 12 years-old and older than 15 years-old Students with uncompleted data at baseline and/or 10-months follow-up Students who dropout the school

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in weekly time in moderate-to-vigorous physical activity at 10 months | baseline and 10-months of intervention
  A list containing 24 types of PA will be used to measure the weekly frequency and the daily duration of each type of PA that the adolescents perform in a typical week.
Change from baseline in the daily time using TV/computer/cellular/video games at 10 months | baseline and 4-months of intervention
  The daily time spent using TV/computer/video games of the individual will be estimated at baseline and after 10 months of intervention.

SECONDARY OUTCOMES:
Change from baseline in the healthy eating score at 10 months | baseline and 10-months of intervention
  Healthy eating score will be estimated using two items related to healthy foods (fruits and vegetables) and three unhealthy (soft drinks, savory and sweets) foods in a typical week. Points from this list will be estimated at baseline and after 10 months of intervention.
Change from baseline in the body mass index at 10 months | baseline and 10-months of intervention
  Body weight (kg) and height (m) will be used to calculate the body mass index (weight/height², kg/m²). Difference between baseline and after 10 months of intervention will be calculated.
Change from baseline in the waist circumference at 10 months | baseline and 10-months of intervention
  Difference in the waist circumference (cm) between baseline and after 10 months of intervention will be calculated.
Change from baseline in the quality of life score at 10 months | baseline and 10-months of intervention
  The quality of life will be measured using the KidScreen instrument. Difference in this score between baseline and after 10 months of intervention will be calculated.
Change from baseline in the sleepiness score at 10 months | baseline and 10-months of intervention
  The difference of frequency and quality of sleep between baseline and after 10 months of intervention will be calculated.
Change from baseline in the academic performance score at 10 months | baseline and 10-months of intervention
  Academic achievement and school attendance will be evaluated in order to create an academic performance score. Difference in this score between baseline and after 10 months of intervention will be calculated.
Change from baseline in the body image score at 10 months | baseline and 10-months of intervention
  The self-assessment of the nine-silhouettes scale proposed by Stunkard et al. will be used to create the body image score. Difference in this score between baseline and after 10 months of intervention will be calculated.

OTHER OUTCOMES:
Change from baseline in the score of intrapersonal PA mediators at 10 months | baseline and 10-months of intervention
  Points obtained from a list of attitude (5 items), expectations (10 items) and self-efficacy (12 items) variables will be estimated at baseline and after 4 months of intervention.
Change from baseline in the score of interpersonal PA mediators at 10 months | baseline and 10-months of intervention
  Points obtained from a list of parental support (7 items), friends support (6 items), physical education teachers (6 items) and general teachers support (6 items) scale will be estimated at baseline and after 4 months of intervention.
Change from baseline in the score of environmental PA mediators at 10 months | baseline and 10-months of intervention
  Points obtained from a list of school environment (4 items) scale will be estimated at baseline and after 10 months of intervention.
Change from baseline in the score of intrapersonal screen time use mediators at 10 months | baseline and 10-months of intervention
  Points obtained from a list of attitude (3 items), expectations (12 items) and self-efficacy (11 items) variables will be estimated at baseline and after 10 months of intervention.
Change from baseline in the score of interpersonal screen time use mediators at 10 months | baseline and 10-months of intervention
  Points obtained from a list of family and friends modelling (4 items), social support (4 items), family beliefs (3 items) and family norms (6 items) variables will be estimated at baseline and after 10 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kelly S Silva, Professor, Principal Investigator — Federal University of Santa Catarina
Locations (1):
- Kelly Samara da Silva, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Costa RM, Lopes MVV, da Costa BGG, Malheiros LEA, Dos Santos PC, Arundell L, da Silva KS. Effect of a school-based multicomponent intervention on time-segmented physical activity and sedentary behavior among adolescents: a cluster randomized control trial. BMC Public Health. 2025 Nov 21;25(1):4090. doi: 10.1186/s12889-025-25314-3. PMID 41272541
- [Derived] da Silva JA, da Silva KS, da Costa BGG, Lopes MVV, Salmon J. Movimente program: effectiveness and moderators of a cluster-randomized controlled trial on self-reported physical activity among Brazilian adolescents. BMC Public Health. 2025 Mar 15;25(1):1017. doi: 10.1186/s12889-025-22130-7. PMID 40089742
- [Derived] Dos Santos PC, Salmon J, Arundell L, Lopes MVV, Silva KS. Effectiveness and moderators of a multicomponent school-based intervention on screen time devices: the Movimente cluster-randomized controlled trial. BMC Public Health. 2021 Oct 13;21(1):1852. doi: 10.1186/s12889-021-11895-2. PMID 34645402
- [Derived] Bandeira ADS, Beets MW, da Silveira PM, Lopes MVV, Barbosa Filho VC, da Costa BGG, Silva KS. Efforts on Changing Lifestyle Behaviors May Not Be Enough to Improve Health-Related Quality of Life Among Adolescents: A Cluster-Randomized Controlled Trial. Front Psychol. 2021 Feb 18;12:614628. doi: 10.3389/fpsyg.2021.614628. eCollection 2021. PMID 33679529
- [Derived] Silva KS, Silva JAD, Barbosa Filho VC, Santos PCD, Silveira PMD, Lopes MVV, Salmon J; "Movimente Program" Working Group. Protocol paper for the Movimente school-based program: A cluster-randomized controlled trial targeting physical activity and sedentary behavior among Brazilian adolescents. Medicine (Baltimore). 2020 Jul 31;99(31):e21233. doi: 10.1097/MD.0000000000021233. PMID 32756101
- [Derived] Knebel MTG, Borgatto AF, Lopes MVV, Dos Santos PC, Matias TS, Narciso FV, Silva KS. Mediating role of screen media use on adolescents' total sleep time: A cluster-randomized controlled trial for physical activity and sedentary behaviour. Child Care Health Dev. 2020 May;46(3):381-389. doi: 10.1111/cch.12755. Epub 2020 Feb 15. PMID 32012323